CLINICAL TRIAL: NCT04071782
Title: Physician Initiated, Prospective, Non-Randomized Single-Center Trial, Investigating the Safety and Efficacy of the Treatment With the Selution Sirolimus Coated Balloon in TASC C and D Tibial Occlusive Disease in Patients With Critical Limb Ischemia From Singapore
Brief Title: Investigating the Safety and Efficacy of the Treatment With the Selution Sirolimus Coated Balloon in TASC C and D Tibial Occlusive Disease in Patients With Critical Limb Ischemia From Singapore
Acronym: PRESTIGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIRB 2019/2121
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Critical Limb Ischemia
Keywords: Angioplasty
MeSH Terms: conditions — Chronic Limb-Threatening Ischemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SELUTION Drug Coated Balloon (Experimental): Study participants will undergo lower limb angioplasty using SELUTION DCB, which is coated with sirolimus.
  Interventions: Device: Drug Coated Balloon

INTERVENTIONS:
Device: Drug Coated Balloon — SELUTION DCB will be used during lower limb angioplasty for treatment of lesions that are TASC C and D, in patients with Critical Limb Ischemia
  Other Names: SELUTION

SUMMARY:
The objective of this clinical investigation is to evaluate the 6-month outcome of the Selution Sirolimus-coated Balloon for the treatment of long tibial occlusive disease (TASC C and D) in patients with Critical Limb Ischemia (CLI)

DETAILED DESCRIPTION:
Extensive arterial occlusion significantly reduces arterial perfusion, and may eventually lead to Critical Limb Ischemia (CLI). The pathology gives rise to symptoms such as ischemic pain, slow healing wounds at lower extremity and gangrene. It places patients with multi-segment occlusion at high risks of amputations and mortality.

The treatment methods for such long occlusive lesions are limited. Traditionally, the standard of care would be surgical revascularization. This is because lesion length have bee identified in several studies as an independent risk factor for the development of restenosis after angioplasty and/or stenting. However, thanks to recent advances in endovascular techniques, such as the utilization of subintimal technique for crossing long segment occlusions, it is now possible to employ endovascular techniques for suitable patients.

The re-establishment of an in-line flow, even if only temporary, can allow tissue healing, which is vital in achieving limb salvage. In addition, the use of Drug Coated Balloons (DCB) and Drug Eluting Stents (DES) can potentially reduce restenosis rate.

To date, there are few studies that have evaluated the performance of DCB in lesions that are longer than 10cm. We hope to evaluate the performance of the Selution DCB when used in treatment of such lesions.

ELIGIBILITY:
Inclusion Criteria:

* Age of subject is > 21 years old
* Patient has Critical Limb Ischemia, presenting a score from 4 to 6 following Rutherford Classification
* Patient is willing to comply with specified follow-up evaluations at the specified times
* Patient understands the nature of the procedure and provides written informed consent, prior to enrolment in the study.
* Patient has a projected life expectancy of at least 12 months and has not suffered an MI within past 30 days
* Prior to enrolment, the guidewire has crossed the target lesion.
* De novo and post-PTA restenotic lesions located in the tibial arteries suitable for endovascular therapy
* Target lesion is located within the native tibial artery
* The length of the target lesion is >100mm and considered as TASC C or D lesion according to the TASC II Classification
* The target lesion has angiographic evidence of stenosis >50% or occlusion, which has been passed with standard guidewire manipulation and predilated to <30% residual stenosis using either POBA or high pressure POBA. No other adjunctive devices have been used to prepare the lesion (example - scoring balloons, rotablator, atherectomy device)
* Target vessel diameter is >1.5mm and <4.5mm below the knee
* Either one or two different tibial arteries may be treated. Lesions in the treated segment may be continuous or may have gaps present between stenoses and occlusions.
* Any tibial vessel intervened on must have distal reconstitution above the ankle
* Inflow iliac, SFA and popliteal lesions can be treated during the same procedure using standard angioplasty and/or approved devices. These inflow lesions must be treated first prior to consideration of treatment of the BTK lesions. The patient can be enrolled if the inflow lesions are treated with good angiographic results (must have <30% residual stenosis and no evidence of embolization)
* There is angiographic evidence of at least one-vessel-runoff through the ankle and into the foot, irrespective of whether or not outflow was re-established by means of previous endovascular intervention.

Exclusion Criteria:

* Patient refusing treatment
* Patient is permanently wheel-chair bound or bedridden
* Presence of a stent in the target lesion that was placed during a previous procedure
* The intervention is being performed in preparation of a planned amputation
* Untreated flow-limiting inflow lesions
* Any previous surgery in the target vessels (including prior ipsilateral crural bypass)
* Previous bypass surgery in the same limb
* Patients for whom antiplatelet therapy, anticoagulants or thrombolytic drugs are contraindicated
* Perforation at the angioplasty site evidenced by extravasation of contrast medium.
* Untreatable lesion located at the distal outflow arteries
* Patients with uncorrectable bleeding disorders
* Aneurysm located at the level of the SFA/popliteal artery
* Non-artherosclerotic disease resulting in occlusion
* Any condition which prevents patients from complying with the study protocol or if patient has a life expectancy of < 1 year.
* Major distal amputation (above the transmetatarsal) in the study limb or non-study limb
* Septicemia or bacteremia
* Patient has undrained pus or spreading wet gangrene in the foot that is not controlled at the time of revascularization procedure
* Neurotrophic ulcer or heel pressure ulcer or ulcer potentially involving calcaneus (index limb)
* Episode of thrombectomy, cutting balloon, lithotripsy, atherectomy or laser devices during procedure
* Any patient considered to be hemodynamically unstable at onset of procedure
* Known allergy to contrast media that cannot be adequately pre-medicated prior to the study procedure
* The patient is currently breast-feeding, pregnant or intends to become pregnant
* Subject receiving immunosuppression therapy, or has known serious immunosuppression therapy, or has known serious immunosuppressive disease (e.g. human immunodeficiency virus), or has severe autoimmune disease that requires chronic immunosuppressive therapy. The patient should also not receive inhibitors of CYP3A (such as Itraconazole, Erythromycin) or inducer of CYP3A (such as Rifampin) within 90 days following procedure
* Patient is participating in another research study of a device, medication, biologic, or other agent within 30 days which could in the opinion of the investigator affect the results of this study
* Patients with lesion to be treated with residual stenosis after POBA of >30%

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2021-01-30 (Actual)

PRIMARY OUTCOMES:
Clinical Primary Safety Endpoint | 30 Days
  Defined as freedom from Major Adverse Event (MAE) - A composite of freedom from device- and procedure-related mortality
Performance Primary Endpoint | 6 Months
  Defined as freedom from clinically driven Target Lesion Revascularization (TLR) within 6 months post-index procedure. Clinically driven TLR is defined as any re-intervention performed for >= 50% diameter stenosis (visual estimate) at the target lesion after documentation of recurrent or unresolved and continuing clinical symptoms of the patient

SECONDARY OUTCOMES:
Primary Patency Rates | 12 Months
  Primary patency defined as absence of a hemodynamically significant stenosis on duplex ultrasound (systolic velocity ratio no greater than 2.5) at the target lesion and without target lesion revascularization within the time of procedure and the given follow-up.
Technical Success | Intra-operative
  Defined as the ability to cross and dilate the lesion and achieve residual angiographic stenosis no greater than 30%
Freedom from clinically-driven TLR | 12 month
  Defined as a repeat intervention to maintain or re-establish patency within the region of the treated arterial vessel plus 5mm proximal and distal to the treated lesion edge at the respective time points
Clinical success at follow-up | 12 months
  Defined as an improvement of Rutherford Classification at all follow-up time points of once class or more as compared to the pre-procedure Rutherford Classification
Wound healing | 6 months
  Defined as closure of primary wound by more than 70% at 6 months or complete healing of primary closed wounds
Freedom from Major Target Limb Amputation | 12 months
Freedom from Severe Adverse Events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Tjun Yip Tang, Principal Investigator — Singapore General Hospital; Tze Tec Chong, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No